CLINICAL TRIAL: NCT00546234
Title: Assessing Treatment Options for Smokers With Asthma.
Brief Title: Tiotropium for Smoking Asthmatics Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No subjects enrolled and no ongoing funding.
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Irvin Mayers, Dr., University of Alberta
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 233372
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2014-08

CONDITIONS: Asthma
Keywords: asthma; tiotropium; smoking; eNO; metabolites; Virtual Asthma Clinic
MeSH Terms: conditions — Asthma; Smoking | interventions — Tiotropium Bromide; Salmeterol Xinafoate; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: tiotropium
- 2 (Active Comparator)
  Interventions: Drug: long acting beta agonist

INTERVENTIONS:
Drug: tiotropium — 18 mcg daily via Handihaler
  Other Names: Spiriva
  Arms: 1
Drug: long acting beta agonist — Turbohaler, 6 & 12 mcg
  Other Names: Serevent; Oxeze
  Arms: 2

SUMMARY:
The study's research questions concern the appropriateness of use of tiotropium for patients with asthma who are current smokers. It is suggested that patients with asthma who smoke, may in fact share similarities with patients with chronic obstructive pulmonary disease (COPD). Because of this, the study will determine whether this sub-group of patients would in fact benefit from therapy currently approved and marketed for COPD patients.

DETAILED DESCRIPTION:
The study is designed as an open label cross-over study. Ethical approval will be obtained from both the University of Alberta Health Research Ethics Board and the University of Saskatchewan Health Research Ethics Board.

Following informed consent, we will obtain pulmonary function testing in all subjects. If subject is currently prescribed a long acting beta agonist (LABA) it will be stopped before continuing with the study and the subject, as with all subjects, will be re-assessed after two weeks. We will also measure exhaled NO (eNO) using standards established by the American Thoracic Society. Additionally we will obtain a urine sample which will be frozen and stored for subsequent metabolite profiling by NMR spectroscopy. Subjects currently prescribed LABA's will have testing done two weeks after stopping medication.

We will obtain routine demographic information including age, sex, and usual asthma medication usage. We will also obtain health related quality of life status using generic (15D) and disease specific (Asthma Quality of Life) questionnaires. Subjects will be instructed regarding use of peak flow meters and the typical symptoms associated with loss of asthma control. They will be instructed regarding accessing a dedicated asthma website (the Virtual Asthma Clinic) that incorporates the above questions. There is also a place for subjects to enter twice daily peak flow measurements. The website is password protected and each subject can access only their own individualized data entry pages. A research coordinator is able to access any subject data again using a unique password. We will use this internet-based program to monitor daily PEF, daily asthma symptoms and asthma-related quality of life. Patients will be instructed to access the website daily and will be re-assessed at two weeks. Subjects will be instructed to continue with their usual asthma management and to log on to the asthma website daily to record symptoms and twice daily peak flows. Peak flows will consist of pre-bronchodilator peak expiratory flow taken in the morning and in the evening. Only subjects meeting criteria for well controlled asthma (GOAL criteria) along with objective compliance with study protocols over the two weeks will then be enrolled in the next phase of the study.

For the next two weeks of the study, subjects will be randomly allocated to take either their regularly prescribed inhaled corticosteroid (ICS) and a long acting beta agonist (LABA) or their regularly prescribed ICS and tiotropium. At the end of this period all subjects will return for spirometry, urine sampling and for measurement eNO. This will be followed by a two week wash-out period when all subjects will take only their inhaled corticosteroid (ICS). For the subsequent two weeks the subject will take the treatment they did not receive in the first two weeks. At the end of this period all subjects will again return for spirometry, urine sampling and for measurement of eNO. During a fifth period of two weeks duration, subjects will take both the LABA and tiotropium. Subjects will then return for final measurement of spirometry, urine sampling and eNO.

Subjects showing variability of symptoms consistent with poor asthma control, will be referred back to their treating physicians with their clinical information. All subjects will be instructed to return to their medication regimen that was initiated by their physician prior to the study.

If subjects experience a clinical exacerbation, they will be instructed to return to their test site. They will be instructed to increase their controller medication and to continue with the increased steroid phase of the study. Any subject experiencing a severe asthma exacerbation (described below) will be withdrawn from the study. Assuming approximately 30% severe exacerbation rate per year in this population, we would anticipate that one to two patients would normally experience a severe exacerbation over a 10 week course. If four of our subjects experience severe exacerbations, we will hold the trial and have an external review of the unblinded data. This will include review of patient compliance with study protocols. If the exacerbations are all in the tiotropium group we will stop the study. We anticipate with the use of the on-line data collection tool (VAC), the study coordinators will be able to see any exacerbation developing at an early point and that we will be able to effectively intervene to prevent severe exacerbations.

A mild clinical exacerbation will be defined by any one of the following events:

1. A decrease in peak flow to less than 80% of best effort for two consecutive days.
2. An increase in reliever medication (fast acting beta agonist) by 50% over baseline needs for two consecutive days.
3. Waking at night due to asthma on two consecutive nights. A severe exacerbation will be defined as any need for additional medical contact for treatment of asthma (e.g., emergency room, walk-in clinic) or any hospital admission for asthma. The need for oral corticosteroids will also constitute a severe exacerbation. If at any point the subjects undergo a severe exacerbation, they will be examined by either their own treating physician or by one of the physicians associated with this study and appropriate escalation of treatment will be commenced. The HREB will be informed of all severe exacerbations. The study coordinator and one of the study physicians will be available by pager during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient with a working diagnosis of asthma by clinical presentation or by spirometry testing results.
* Currently prescribed inhaled corticosteroids (ICS) for the treatment of asthma, and may or may not be prescribed additional therapies for asthma.
* Is a current smoker with a minimum of a five year history of smoking.
* Provides written informed consent.

Exclusion Criteria:

* Has a diagnosis of COPD.
* Is currently enrolled in another clinical trial.
* Has any condition which, may decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
* Is unable to provide written informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To evaluate whether current smokers with asthma benefit from the introduction of tiotropium. | 10 weeks

SECONDARY OUTCOMES:
To assess whether there are specific genotypes that identify specific asthma patient populations that may benefit from this therapy. | 10 weeks
To determine if the Virtual Asthma Clinic is an acceptable tool for data collection in a clinical trial setting. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Irvin Mayers, MD, FRCPC, Principal Investigator — University of Alberta; Darcy Marciniuk, MD, Principal Investigator — University of Saskatchewan; Dilini Vethanayagam, MD, Principal Investigator — University of Alberta; Harissios Vliagoftis, MD, Principal Investigator — Unviersity of Alberta
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal University Hospital, Saskatoon, Saskatchewan